CLINICAL TRIAL: NCT06455488
Title: MANAGEment of Ventricular Tachycardia Outcomes Registry
Brief Title: MANAGE-VT Registry - MANAGEment of Ventricular Tachycardia Outcomes Registry
Acronym: MANAGE-VT
Status: Recruiting | Type: Observational
Sponsor: CorVita Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-CSF-00300
Record Dates: First submitted 2024-06-05; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Ventricular Tachycardia
Keywords: ventricular arrhythmia; ventricular tachycardia; ventricular fibrillation; stroke
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Stroke | interventions — Defibrillators, Implantable; Anti-Arrhythmia Agents; Anticoagulants; Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- MANAGE-VT Patients: Patients will be assessed on the status of their ventricular tachycardia as well as other criteria such as: EKG,
  Interventions: Procedure: Ventricular Tachycardia Ablation; Device: ICD Implant; Drug: Antiarrhythmic drug; Diagnostic Test: EKG; Diagnostic Test: Cardioversion; Diagnostic Test: Echocardiogram

INTERVENTIONS:
Procedure: Ventricular Tachycardia Ablation — This is a surgical ablation meant to reset patients irregular rhythm back to sinus.
Device: ICD Implant — A pacemaker or defibrillator implant to prevent SCD
  Other Names: Pacemaker Implant
Drug: Antiarrhythmic drug — Drug therapies
  Other Names: Statin Therapy; Anticoagulants
Diagnostic Test: EKG — Monitoring EKG testing done on registry patients
Diagnostic Test: Cardioversion — Monitoring cardioversions on registry patients
Diagnostic Test: Echocardiogram — Monitoring echocardiogram testing done on patients

SUMMARY:
Data collection registry for patients with ventricular tachycardia to help physicians give better care for patients clinically and procedurally.

DETAILED DESCRIPTION:
After consent from a patient the research team will input patients data from many different categories. There is a link to the PDF for the consent form, a patients anticoagulant medications will be assessed, their ventricular tachycardia (VT) history will be inputted, and their date of birth and zip code will inputted. The research team will then input any EKG's, echocardiograms, VT ablations, ICD's, S-ICD's, lab results, and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old
* Must not be

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who have been diagnosed and have evidence of ventricular tachycardia and are over the age of 18. Every patient was presented with a consent form and was given a description of the study in a clinical setting.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2030-07-20 (Estimated); Study Completion 2030-07-20 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Ventricular Tachycardia | July 20, 2020 - Present
  The natural progression of v-tach will be assessed through medical record review
Number of Participants with Risk of Sudden Cardiac Death | July 20, 2020 - Present
  All events of sudden cardiac death that arise from patients with ventricular tachycardia
Prevent Risk of Stroke | July 20, 2020 - Present
  All strokes, transient ischemic and systemic thrombo-embolic events

CONTACTS AND LOCATIONS:
Locations (1):
- Corvita Science Foundation, Chicago, Illinois, United States